CLINICAL TRIAL: NCT04757844
Title: The Effects of Different Attentional Focus During Walking on Prefrontal Cortical Activation in Young Healthy Adults
Brief Title: Attentional Focus and Prefrontal Cortical Activation
Acronym: AttNIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO 2020-22
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: near infrared spectroscopy; prefrontal cortex; attention; gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young healthy voluntary adults (Experimental): 30 young healthy voluntary adults
  Interventions: Device: Functional Near-Infrared Spectroscopy (fNIRS)

INTERVENTIONS:
Device: Functional Near-Infrared Spectroscopy (fNIRS) — The hemodynamic response in prefrontal cortex will be measured using an Octamon+ system (Artinis). Eight emission and two detector probes will be arranged on the participant's forehead.

SUMMARY:
Attention may influence the motor performance and frontal activity. This study will examine the effect of different attentional focus : internal, external and divided attention (dual task) on prefrontal cortical activation (fNIRS) and on gait performance. Thirty young healthy voluntary adults will participate in this study.

DETAILED DESCRIPTION:
The subjects will be guided to walk at a normal pace while maintaining the required attentional focus. They will walk on 30 m five times in each of the four different focus conditions :1) no instructions about the attentional focus 2) internal focus on their feet movements, 3) external focus on two lines drawn on the floor, 4) divided attention (walking while performing an arithmetic task). A fNIRS system will be used for the prefrontal cortex activation evaluation and FeetMe soles for gait analyses.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* 18 -30 years old
* Informed consent obtained
* Free from any neurological, cardiologic, rheumatologic disorders.

Exclusion Criteria:

* Assisted walker.
* Disorders affecting gait.
* Concomitant medication likely to interfere with the results.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Effects of different attentional conditions on hemodynamic response in prefrontal cortex | Baseline
  Oxyhemoglobin variations in prefrontal cortex measured with fNIRS
Effects of different attentional conditions on hemodynamic response in prefrontal cortex | Baseline
  Deoxyhemoglobin variations in prefrontal cortex measured with fNIRS

SECONDARY OUTCOMES:
Effects of speed on gait. | Baseline
  Gait parameters will be measured with connected soles FeetMe ® : speed
Effects of cadence on gait. | Baseline
  Gait parameters will be measured with connected soles FeetMe ® : cadence
Effects of stride length on gait. | Baseline
  Gait parameters will be measured with connected soles FeetMe ® : stride length
Effects of double support time on gait. | Baseline
  Gait parameters will be measured with connected soles FeetMe ® : double support time

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wulf G, Hoss M, Prinz W. Instructions for motor learning: differential effects of internal versus external focus of attention. J Mot Behav. 1998 Jun;30(2):169-79. doi: 10.1080/00222899809601334. PMID 20037032
- [Background] Kim SA, Ryu YU, Shin HK. The effects of different attentional focus on poststroke gait. J Exerc Rehabil. 2019 Aug 28;15(4):592-596. doi: 10.12965/jer.1938360.180. eCollection 2019 Aug. PMID 31523682
- [Background] Lu CF, Liu YC, Yang YR, Wu YT, Wang RY. Maintaining Gait Performance by Cortical Activation during Dual-Task Interference: A Functional Near-Infrared Spectroscopy Study. PLoS One. 2015 Jun 16;10(6):e0129390. doi: 10.1371/journal.pone.0129390. eCollection 2015. PMID 26079605
- [Background] Herold F, Wiegel P, Scholkmann F, Thiers A, Hamacher D, Schega L. Functional near-infrared spectroscopy in movement science: a systematic review on cortical activity in postural and walking tasks. Neurophotonics. 2017 Oct;4(4):041403. doi: 10.1117/1.NPh.4.4.041403. Epub 2017 Aug 1. PMID 28924563
- [Background] Farid L, Jacobs D, Do Santos J, Simon O, Gracies JM, Hutin E. FeetMe(R) Monitor-connected insoles are a valid and reliable alternative for the evaluation of gait speed after stroke. Top Stroke Rehabil. 2021 Mar;28(2):127-134. doi: 10.1080/10749357.2020.1792717. Epub 2020 Jul 13. PMID 32654627
- [Background] Kal EC, van der Kamp J, Houdijk H. External attentional focus enhances movement automatization: a comprehensive test of the constrained action hypothesis. Hum Mov Sci. 2013 Aug;32(4):527-39. doi: 10.1016/j.humov.2013.04.001. Epub 2013 Jun 30. PMID 24054892
- [Background] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Background] Wood JN, Grafman J. Human prefrontal cortex: processing and representational perspectives. Nat Rev Neurosci. 2003 Feb;4(2):139-47. doi: 10.1038/nrn1033. No abstract available. PMID 12563285
- [Background] Pelicioni PHS, Tijsma M, Lord SR, Menant J. Prefrontal cortical activation measured by fNIRS during walking: effects of age, disease and secondary task. PeerJ. 2019 May 3;7:e6833. doi: 10.7717/peerj.6833. eCollection 2019. PMID 31110922
- [Background] Shafizadeh M, Platt GK, Mohammadi B. Effects of different focus of attention rehabilitative training on gait performance in Multiple Sclerosis patients. J Bodyw Mov Ther. 2013 Jan;17(1):28-34. doi: 10.1016/j.jbmt.2012.04.005. Epub 2012 May 10. PMID 23294680
- [Background] Yogev-Seligmann G, Rotem-Galili Y, Mirelman A, Dickstein R, Giladi N, Hausdorff JM. How does explicit prioritization alter walking during dual-task performance? Effects of age and sex on gait speed and variability. Phys Ther. 2010 Feb;90(2):177-86. doi: 10.2522/ptj.20090043. Epub 2009 Dec 18. PMID 20023000
- [Background] Holtzer R, Mahoney JR, Izzetoglu M, Izzetoglu K, Onaral B, Verghese J. fNIRS study of walking and walking while talking in young and old individuals. J Gerontol A Biol Sci Med Sci. 2011 Aug;66(8):879-87. doi: 10.1093/gerona/glr068. Epub 2011 May 17. PMID 21593013
- [Background] Udina C, Avtzi S, Durduran T, Holtzer R, Rosso AL, Castellano-Tejedor C, Perez LM, Soto-Bagaria L, Inzitari M. Functional Near-Infrared Spectroscopy to Study Cerebral Hemodynamics in Older Adults During Cognitive and Motor Tasks: A Review. Front Aging Neurosci. 2020 Jan 21;11:367. doi: 10.3389/fnagi.2019.00367. eCollection 2019. PMID 32038224